CLINICAL TRIAL: NCT02966418
Title: The Effects of Intermittent Whole-body Hypoxic Preconditioning on Patients With Carotid Artery Stenosis
Brief Title: Hypoxic Preconditioning on Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hua Yan (Other)
Responsible Party: Sponsor-Investigator, Hua Yan, Director, Tianjin Huanhu Hospital
Organization: Tianjin Huanhu Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JH2016-17
Record Dates: First submitted 2016-11-06; First posted 2016-11-17 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Hypoxic Preconditioning; Carotid Artery Stenosis; Ischemic Cerebrovascular Disease
Keywords: Hypoxic preconditioning; Carotid artery stenosis; Ischemic cerebrovascular disease
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild hypoxia preconditioning (Active Comparator): Patients will be treated with mild hypoxia (Note: The oxygen concentration decreased from 20% to 18%, and keeping at 18%) before surgery.
  Interventions: Procedure: Mild Hypoxia Preconditioning
- Sham preconditioning (Sham Comparator): Patients will be treated with sham preconditioning (oxygen concentration: 21％) before surgery.
  Interventions: Procedure: Sham preconditioning

INTERVENTIONS:
Procedure: Mild Hypoxia Preconditioning — Patients will be treated with mild hypoxia ( Note: The oxygen concentration decreased from 20% to 18%, and keeping at 18%)×7 days，twice a day in the morning and in the afternoon before surgery.
  Arms: Mild hypoxia preconditioning
Procedure: Sham preconditioning — Patients will be treated with sham preconditioning (oxygen concentration: 21％) ×7 days，twice a day in the morning and in the afternoon before surgery.
  Arms: Sham preconditioning

SUMMARY:
The purpose of this study is to study the effects of intermittent whole-body hypoxic preconditioning on patients with carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Informed written consent from the patient.
2. Han nationality, age >18 years.
3. Carotid artery stenosis on at least one side, measuring more than 70% by ultrasonic detection and requiring carotid artery stenting or a carotid endarterectomy.
4. Long-term residence at an altitude of <100 m (the altitude of Tianjin is 2-5 m).
5. Not having been to an altitude ≥1500 m in two years.

Exclusion Criteria:

1. Planned vessel sacrifice as the primary modality for ischemic cerebrovascular treatment.
2. Systemic blood disease before intervention.
3. Regular physical activity exercise: frequency >1 time/week, duration >20 min.
4. History of brain disease or history of stroke or transient ischemic attack within the previous six months.
5. History of heart, liver, kidney or lung disease.
6. History of hypertension and poor blood pressure control, with blood pressure >160/90 mmHg.
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | Before, during and 5 min after the intervention.
Heart rate | Before, during and 5 min after the intervention.
Systolic blood pressure | Before, during and 5 min after the intervention.
Arterial blood oxygen saturation | Before, during and 5 min after the intervention.
Hemoglobin content | On admission, and at the 1st day after surgery.
Hypoxia inducible factor-1α | On admission, and at the 1st day after surgery.
Erythropoietin | On admission, and at the 1st day after surgery.
Vascular endothelial growth factor | On admission, and at the 1st day after surgery.
Neuron-specific enolase | On admission, and at the 1st day after surgery.
S100β protein | On admission, and at the 1st day after surgery.
Brain-derived neurotrophic factor | On admission, and at the 1st day after surgery.

SECONDARY OUTCOMES:
Serum aspartate transaminase | On admission, and at the 1st day after surgery.
Serum alanine aminotransferase | On admission, and at the 1st day after surgery.
Serum creatinine | On admission, and at the 1st day after surgery.
Blood urea nitrogen | On admission, and at the 1st day after surgery.
The incidence of adverse events | During the intervention.
Average length of hospital stay | Through study completion, an average of 3 months.
Postoperative complications | Through study completion, an average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Yan, Doctor, Study Chair — Tianjin Huanhu Hospital
Locations (1):
- Tianjin HuanHu Hospital, Tianjin, Tianjin Municipality, China